CLINICAL TRIAL: NCT03706092
Title: Impact of the Intervention of Pharmacists and Geriatrician on Drug Prescription in Critically Ill Elderly Patients Admitted in Surgical ICU
Brief Title: Impact of the Intervention of Pharmacists and Geriatrician on Drug Prescription in Elderly Patients in a Surgical ICU
Acronym: IATROAGE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: IATROAGE
Record Dates: First submitted 2018-08-16; First posted 2018-10-15 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2019-12

CONDITIONS: Aged; Critical Care
Keywords: iatrogenic; surgery ICU; quality of life; disability; inappropriate medications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before: Elderly patients > = 70 in ICU without any intervention of the pharmacists and of the geriatricians
- After: Elderly patients > = 70 in ICU with individualized intervention of the pharmacists and of the geriatricians

SUMMARY:
In order to optimize drug prescription and to reduce potentially inappropriate medications, a pharmaceutical analysis activity is conducted in our establishment for several years. Medical prescriptions are reviewed daily by pharmacists. This activity is developed in approximatively 84% of the hospital wards of the institution, and especially in the geriatric department. Drug induced adverse effects are frequently encountered in elderly people and ICU environment causes a high risk of iatrogenic events because of the complexity of care and of the severity of illness. The hypothesis of the study is that the intervention of pharmacists and geriatricians could improve the medical prescription in elderly patients by reducing avoidable drug interactions and thus by decreasing the risk of drug induced adverse effects.

The primary objective of this study is to evaluate the impact of the intervention of pharmacists and geriatricians on medical prescription and on iatrogenic risk in elderly critically ill patients admitted in surgical ICU. The secondary objectives are (i) to describe the elderly patients population in surgical ICU, (ii) to analyze the impact of the ICU stay on medical prescription, (iii) to analyze the opportunities suggested by the pharmacists to optimize drug therapies and (iv) to assess the impact of drug prescription in the ICU on long-term disability.

A prospective, observational, before-after study will be conducted from august 1, 2018 to February 1, 2020, in the surgical ICU of the hospital. Patients older than 70 years and admitted to surgical ICU will be eligible. This study will be conducted in 2 successive steps: (1) first step: without any intervention of pharmacists or and geriatricians (Baseline), (2) second step: all drug prescription during the ICU and the hospital stay will be analyzed by a pharmacist and a geriatrician, to decrease drug interaction and risk of drug related adverse effect. During each step, the demographic and medical data will be recorded. Medical prescriptions will be reviewed at ICU admission, at 96 hours after ICU admission and then every 4 days until discharge from the ICU. For each patient, the impact of the intervention on mid-term and long-term disability will be assessed during a geriatric evaluation by using adequate specific scale at hospital discharge and at 3 months after hospital discharge. All iatrogenic events will be collected and analyzed.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the impact of the intervention of pharmacists and geriatricians on medical prescription and on the iatrogenic risk in elderly critically ill patients admitted in surgical ICU. This study is before-after prospective study, carried out in 2 steps.

Step 1 data collection from August 1, 2018 to February 1, 2019

This step is a prospective analysis without any intervention of the pharmacist and of the geriatrician.

* The sociodemographic, and medical (comorbidities, reason for ICU admission, SAPS II (Simplified Acute Physiology Score) and SOFA (Sepsis-related Organ Failure Assessment) scores, laboratory data, invasive procedures data will be collected from ICU medical record.
* A geriatric evaluation and disability evaluation will be performed by using the ADL (Activity of Daily Living), Charlson, and SEGA (Short Emergency Geriatric Assessment) scales.
* The medical prescriptions will be reviewed at the first day and at 96 hours after admission in the ICU, and every 4 days during ICU stay. The pharmacist will analyse the medical prescriptions by using a standardized tool (Micromedex®, Theriaque®, Vidal®), to identify inappropriate prescription, and to assess the iatrogenic risks. These interventions will be quantified by using the SFPC Scale (French Society of clinical pharmacy).
* Iatrogenic events will be reported and analyzed.
* Drug prescription and patient outcome at discharge from the ICU and at discharge from the hospital will be collected.
* At 3 months from discharge from the hospital, a new geriatric evaluation will be conducted (patient's outcome and medical prescription).

Step 2, from March 1, 2019 to March, 2020.

This step is a prospective analysis with the intervention of the pharmacist and of the geriatrician.

The same data that step 1 will be collected. During this step, the pharmacist carries individualized interventions that will be discuss with the physician in charge of the patient to improve the safety of drug prescription. The physician will be allowed to accept or to refuse these interventions.

At 3 months from discharge from the hospital, a consultation with geriatrician will be proposed to the elderly patient. The geriatric evaluation and disability assessment will be conducted during this consultation.

ELIGIBILITY:
Inclusion Criteria:

* patients 70 years or older
* admitted to surgical ICU

Exclusion Criteria:

* patients refusing data collection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 70 years or older patient admitted to surgical ICU of university affiliated hospital of Besançon
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Impact of geriatric and pharmacist's intervention | Hospital stay until 3 months after
  Difference between iatrogenic risks before/after pharmaceutical intervention on the elderly's prescription. The iatrogenic risk is evaluated with the iatrogenic events rates and the inappropriate prescriptions rates.

SECONDARY OUTCOMES:
Describe the medical characteristics of elderly patients population in surgical intensive care with the Charlson Comorbidities Index (CCI) | During hospital stay up to 3 months after discharge
  Charlson Comorbidities Index
  Three grades of severity:
  mild, with CCI scores of 1-2; moderate, with CCI scores of 3-4; severe, with CCI scores ≥5
Describe the medical characteristics of elderly patients population in surgical intensive care | During hospital stay up to 3 months after discharge
  Rates of hospitalization's causes: surgical emergency causes, elective surgery causes, medical emergency causes, elective medical causes
Describe the demographic elderly patients population in surgical intensive care | During hospital stay up to 3 months after discharge
  age, sex
Impact of a stay surgical intensive care on medical prescription change | During Hospital stay in ICU (Day 0, 4, 8, 12, 16) and 3 months after discharge
  number of new treatment, number of new interaction, number of iatrogenic event, before/after surgical intensive care
Evaluate the intervention's impact on the disability and geriatric evaluation with ADL scale | 3 months after hospital discharge
  Evolution of disability and geriatric evaluation before/after intervention:
  - ADL (Activity Daily Living evolution of the different geriatrics scores) 0 : dependance, 6 autonomy
Evaluate the intervention's impact on the disability and geriatric evaluation with SEGA scale | 3 months after hospital discharge
  Evolution of disability and geriatric evaluation before/after intervention:
  - SEGA (Short Emergency Geriatric Assessment): 0-26 < or = 8 : Low fragility, 9-11: fragility, > or = 12 Very fragile person
Analyse the opportunities suggested by the pharmacist for optimization of drug therapies | During Hospital stay ICU (Day 0, 4, 8, 12, 16)
  rates of kind opportunities suggested by the pharmacist (dosage adjustment, galenic form change, inappropriate medication ...)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Laure CLAIRET, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France